CLINICAL TRIAL: NCT05575830
Title: Immune Response to the Recombinant Zoster Vaccine in People Living With HIV Over 50 Years of Age Compared to Non-HIV Age- and Gender-matched Controls - The Shingr'HIV Phase IV Multicenter Study
Brief Title: Immune Response of Shingrix Vaccine in People Living With HIV (> 50 y.o.) Compared to Age-matched Controls
Acronym: Shingr'HIV
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Calmy Alexandra (Other)
Responsible Party: Sponsor-Investigator, Calmy Alexandra, Prof, University Hospital, Geneva
Organization: University Hospital, Geneva (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2022-01314; 2023-504482-23 (EudraCT Number)
Record Dates: First submitted 2022-09-01; First posted 2022-10-12 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-08

CONDITIONS: RZV Vaccine (Shingrix ®)
Keywords: RZV vaccine; PLWH; Immune response; Safety

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- RZV or Shingrix®) (Experimental): Recombinant Zoster Vaccine
  Interventions: Biological: Recombinant Zoster Vaccine

INTERVENTIONS:
Biological: Recombinant Zoster Vaccine — Shingrix® vaccine will be administered in two vaccinations on Day0 and Day60
  Other Names: (Shingrix® )

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of the adjuvanted recombinant Zoster vaccine (RZV, or Shingrix®) in older people (> 50 years) living with HIV (PLWH) compared to age-matched healthy adults over a 1-year period.

DETAILED DESCRIPTION:
This is a prospective multicentric phase IV study, aiming at evaluating the immunogenicity and safety profile of RZV in PLWH over 50 years of age (YOA) on long term antiretroviral therapy (ART) (>10 years) compared to non-HIV age-matched adult controls to address the combined effect of aging and immunosuppression from HIV disease.

Inclusion will be stratified as follow:

HIV+ groups:

* Group 1: PLWH registered in the SHCS or ANRS CO3, >75 YOA and under cART for more than 10 years - N=50
* Group 2: PLWH patients registered in the SHCS, aged between 60 and 75 and under cART for more than 10 years - N=50
* Group 3: PLWH patients registered in the SHCS, aged between 50 and 59 and under cART for more than 10 years - N=50

Control groups:

* Group 4: Healthy adults aged >75 YOA- N=25
* Group 5: Healthy adults aged between 60 and 75 - N=25
* Group 6: Healthy adults aged between 50 and 59 - N=25

In addition, participants of all groups will be proposed to be included in the "Innate substudy" (target of 15 participants/group) and have two additional blood drawings 1 day after each vaccine dose to measure innate response triggered by RZV.

Participants will receive Shingrix® on Day0 and Day60; immunological response will be assessed on Day 1, Day61, Day90, Day360.

Unsolicited Adverse events of special intesrest (AESI) will be collected on Day 28, Day 60, Day90, Day360; patients reported outcomes (PROs) will be declared for one week after each vaccination.

ELIGIBILITY:
Inclusion Criteria:

For PLWH:

* Be registered in the SHCS or in the ANRS CO3 Aquitaine Cohort
* Age >50 YOA
* Time since cART initiation > 10 years
* Not already vaccinated with RZV
* HIV viral load <50 copies/ml (within 6 months from the last blood sampling)
* Informed consent as documented by signature
* (France) : Person affiliated with or beneficiary of the French social security scheme

For aged/gender-matched controls

* Age >50 YOA
* Not already vaccinated with RZV
* Informed consent as documented by signature
* (France) Not HIV infected
* (France) Person affiliated with or beneficiary of the French social security scheme

Exclusion Criteria:

* Ongoing signs of febrile or non-febrile infection at the time of the first vaccination
* Immunosuppression from the following:

  * Current malignant neoplasm;
  * primary immunodeficiency;
  * recent (<2 years) solid or bone-marrow transplant or any transplant still requiring immunosuppressive therapy
* Intake of drugs which suppress the immune system (e.g. glucocorticoids for a long time [an equivalent dose of prednisolone >20 mg/day > 3 months], monoclonal antibodies, cytostatics, biological products, etc.) within 6 months before screening.
* Administration of immunoglobulins or any blood products within 3 months preceding the first dose of vaccine or planned administration during the study period
* Having received a vaccine in the last month or is expected to receive a vaccine in the next month
* Having received a shingles vaccine within one year
* Presented with herpes zoster in the previous year
* Contra-indication to RZV
* Hospitalized patients
* Unable to provide informed consent or inability to follow the procedures of the study, e.g. due to language problems, psychological disorders, dementia, etc. of the participant
* Participation in another study with investigational drug within the 30 days preceding and during the present study.
* (France) Pregnant or breastfeeding woman
* (France) Patient governed by articles L 1121-5 to L 1121-8 (persons deprived of their liberty by a judicial or administrative decision, minors, persons of legal age who are the object of a legal protection measure or unable to express their consent)

Ages: 50 Years to 95 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 225 (Estimated)
Dates: Start 2022-12-14 (Actual); Primary Completion 2025-04-16 (Actual); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Geometric mean titer (GMT) of gE-specific total IgG | Day 90
  gE-specific total IgG titers is determined by gE-specific ELISA from sera samples

SECONDARY OUTCOMES:
Vaccine safety - AESI 7 days | 7 days
  Incidence adverse events of special interest (AESI) in the 7 days following each vaccination (reactogenicity) collected in a diary card
Vaccine safety - SAE 360 days | 360 days
  Incidence of SAE throughout the study period
Vaccine safety -pIMDs | 360 days
  Incidence of potential immune mediated disorders (pIMDs) throughout the study period
Vaccine safety - PLWH | Day 90
  In PLWH: Percentage of PLWH with viral load >50 copies/ml one month after the second RZV vaccination (D90)
Vaccine immunogenicity - CD4+ T cells | Day 90
  Mean of gE-specific CD4+ T cells expressing at least 2 activation markers (i.e. CD40L, IFN-gamma, IL-2 or TNF-alpha) per million of T cells, measured at D90

CONTACTS AND LOCATIONS:
Overall Officials: Alexandra Calmy, Prof. MD, Study Director — University Hospitals of Geneva, Infectious disease department,
Locations (10):
- France (3):
  - Hôpital Saint-André, CHU de Bordeaux, Bordeaux, Bordeaux
  - SMIT - Service de Maladies Infectieuses et Tropicales Le Tripode -Groupe Hospitalier Pellegrin, Bordeaux, France
  - CHU de Bordeaux - Hôpital Haut-Lévèque, Pessac, Gironde
- Switzerland (7):
  - University Hospital Basel, Basel, Basel
  - Bern University Hospital (Inselspital), Bern, Canton of Bern
  - University Hospitals of Geneva, Geneva, Canton of Geneva
  - Kantonsspital, Sankt Gallen, Canton of St. Gallen
  - Centre Hospitalier Universitaire Vaudoise (CHUV), Lausanne, Canton of Vaud
  - University Hospital Zurich, Zurich, Canton of Zurich
  - Ente Ospedaliero Cantonale, Lugano, Canton Ticino

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hentzien M, Bonnet F, Bernasconi E, Biver E, Braun DL, Munting A, Leuzinger K, Leleux O, Musardo S, Prendki V, Schmid P, Staehelin C, Stoeckle M, Walti CS, Wittkop L, Appay V, Didierlaurent AM, Calmy A. Immune response to the recombinant herpes zoster vaccine in people living with HIV over 50 years of age compared to non-HIV age-/gender-matched controls (SHINGR'HIV): a multicenter, international, non-randomized clinical trial study protocol. BMC Infect Dis. 2024 Mar 19;24(1):329. doi: 10.1186/s12879-024-09192-5. PMID 38504173
- See also: Shingrix vaccine information — https://www.ema.europa.eu/documents/product-information/shingrix-epar-product-information_en.pdf